CLINICAL TRIAL: NCT01950650
Title: GAPP 1 Survey: Global Attitudes of Patients and Physicians in Insulin Therapy for Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GAPP1; U1111-1136-2507 (Other: WHO)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with diabetes
  Interventions: Behavioral: No treatment given
- Physicians
  Interventions: Behavioral: survey

INTERVENTIONS:
Behavioral: No treatment given — Survey conducted through computer-assisted telephone interviewing.
  Groups: Patients with diabetes
Behavioral: survey — Survey conducted via the Internet.
  Groups: Physicians

SUMMARY:
This study is conducted in Asia, Europe and in the United States of America. The aim of this study is to examine patient and physician beliefs regarding insulin therapy and the degree to which patients adhere to their insulin regimens.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS WITH DIABETES:
* Age 18 years or older
* Treated with insulin
* Type 1 or Type 2 diabetes
* PHYSICIANS:
* In practice for more than 1 year since completing residency
* See a minimum number of patients with diabetes per week (primary care physicians 5, specialists 10)
* Initiate insulin treatment for patients with diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Insulin treated patients with diabetes (type 1 or 2), and physicians involved in the treatment, management of diabetes and care of patients with diabetes.
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Frequency of insulin omission/non-adherence | In the past 30 days prior to the day when responding to the survey (patient survey)
Reasons for insulin omission/non-adherence reported by patient and physician | Day 1 (when responding to the survey)

SECONDARY OUTCOMES:
Impact of insulin treatment on life domains (patient survey) | Day 1 (when responding to the online questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (10):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Bangalore, India
- Novo Nordisk Investigational Site, Tokyo, Japan
- Novo Nordisk Investigational Site, Moscow, Russia
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- [Result] Peyrot M, Barnett AH, Meneghini LF, Schumm-Draeger PM. Insulin adherence behaviours and barriers in the multinational Global Attitudes of Patients and Physicians in Insulin Therapy study. Diabet Med. 2012 May;29(5):682-9. doi: 10.1111/j.1464-5491.2012.03605.x. PMID 22313123
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com